CLINICAL TRIAL: NCT03856229
Title: Shortened Steroid Therapy in Patients With Moderate and Severe Pneumonia Due to P. Jirovecii Associated With HIV / AIDS
Brief Title: Short-term Steroid Therapy in Patients With P. Jirovecii Pneumonia Due to HIV / AIDS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Investigación en. Enfermedades Infecciosas, Mexico (Other Government)
Responsible Party: Principal Investigator, Gustavo Reyes-Teran, Principal Investigator, Centro de Investigación en. Enfermedades Infecciosas, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C40-18
Record Dates: First submitted 2019-02-08; First posted 2019-02-27 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Pneumocystis; HIV/AIDS; Steroid
Keywords: HIV/AIDS; PCP treatment; Steroids for PCP
MeSH Terms: conditions — Pneumonia, Pneumocystis; Acquired Immunodeficiency Syndrome | interventions — Costs and Cost Analysis

STUDY DESIGN:
Intervention Model Description: After obtaining the informed consent. The subjects will be randomized 6 days after starting treatment for PCP with trimethoprim/ sulfamethoxazole plus prednisone or methylprednisolone. Stratified randomization will be generated by an electronic system, in blocks of 6 and 8, and a 1:1 ratio, according to the CD4+ T cell count (less or more than 50 cells/mm3 and assigned to each group:
  * Group A or Conventional Steroids use (CoSt). Patients will receive 21 days of steroid treatment.
  * Group B or Shortened Steroids use (SSt). Subjects with moderate PCP will receive 8 days of steroids and subjects with severe PCP 14 days of steroids.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A conventional steroid regimen (Active Comparator): Subjects will receive the conventional steroid regimen with prednisolone or equivalent (with methylprednisolone): Day 1 to 5: 40 mg orally every 12 h; Day 6 to 10: 40 orally every 24 hours; and Day 11 to 21: 20 mg orally every 24 h.
  Interventions: Drug: Conventional steroid regimen
- Group B shortened steroid regimen (Experimental): Subjects will receive the shortened steroid regimen for the severity of pneumonia with prednisone or equivalent with methylprednisolone, depending the severity of pneumonia:
  * Moderate PCP. 40 mg orally every 12 h (Day 1 to 5);40 mg orally every 24 hours (Day 6 to 8).
  * Severe PCP. 40 mg orally every 12 h (Day 1 to 5),40 mg orally every 24 hours (Day 6 to 10); and 20 mg orally every 24 h (Day 11 to 14).
  Interventions: Drug: Shortened steroid regimen

INTERVENTIONS:
Drug: Conventional steroid regimen — Subjects will receive the conventional steroid regimen with prednisolone or equivalent (with methylprednisolone): Day 1 to 5: 40 mg orally every 12 h; Day 6 to 10: 40 orally every 24 hours; and Day 11 to 21: 20 mg orally every 24 h.
  Other Names: CoSt
  Arms: Group A conventional steroid regimen
Drug: Shortened steroid regimen — * Subjects with Moderate PCP. Prednisolone (or equivalent with methylprednisolone) 40 mg orally every 12 h (Day 1 to 5);40 mg orally every 24 hours (Day 6 to 8).
  * Subjects with severe PCP. Prednisolone (or equivalent with methylprednisolone) 40 mg orally every 12 h (Day 1 to 5),40 mg orally every 24 hours (Day 6 to 10); and 20 mg orally every 24 h (Day 11 to 14).
  Other Names: SSt
  Arms: Group B shortened steroid regimen

SUMMARY:
The treatment guidelines for Pneumocystis pneumonia (PCP) suggest adding 40mg of prednisone (or its equivalent in methylprednisolone) twice per day on days 1 through 5, 40 mg days 6 through 10, and 20 mg daily on days 11 through 21 in subjects with moderate and serious PCP. Steroids have shown to improve clinical outcome and reduction in mortality in HIV-infected patients the effectiveness of adjuvant steroid treatment for PCP has been observed if it starts within the first 24 to 48 hours. Possibly, there is a long-term benefit with their use in the recovery of function and limitation of chronic pulmonary complications; recently, benefits have been observed in decreasing the incidence of Inflammatory Immune Reconstitution Syndrome (IRIS) due to Mycobacterium tuberculosis. On the other hand, steroids could increase the morbidity related to adverse reactions as well as paradoxical worsening of associated herpes virus infection, which are attributed to IRIS or as a result of immunosuppression generated by their use. Recently, it has been shown that gradually steroids withdrawal is not necessary in patients who have received less than 21 days of treatment.

This non-inferiority work aims to confirm the null hypothesis that a reduced steroid scheme in patients with moderate PCP (8 days) and severe pneumonia (14 days) is sufficient to limit long-term ventilatory complications and acute postinflammatory syndrome, compared to the conventional 21-day scheme. It also has been hypothesized that it could be associated with fewer cases of IRIS due to herpes virus type 1,2,3 and 8.

DETAILED DESCRIPTION:
The investigators selected hospitalized subjects with confirmed or suspected moderate or severe PCP: the diagnostic certainty will be based on the following criteria:

Proved PCP. Defined as cases with presence of P. jirovecii cysts in bronchial alveolar lavage (BAL) exams or lung biopsy.

Possible PCP. Defined by the following two criteria: 1) the presence of three of four items: cough, fever, dyspnea and compatible radiological or tomographic findings 2) associated clinical improvement after the onset of trimethoprim/sulfamethoxazole (TMP / SMX).

Probable PCP. Defined as the presence of one of the two previous criteria, without other identified microorganisms.

The radiological or tomographic findings compatible with PCP are: presence of bilateral reticular infiltrate, ground glass, crazy paving pattern and presence of bullae, cysts or spontaneous pneumothorax.

The microbiological findings will be the identification of cysts in the Grocott stain or a positive immunofluorescence test (IFA).

Patients will be classified as moderate PCP when the partial pressure of oxygen (PaO2) is less than 70 mmHg and the alveolar arterial difference (Da-a) is greater than 35 mmHg and severe PCP when it is greater than 45 mmHg.

The sample size was calculated for non-inferiority tests to a tail with an estimated mortality of 16% for both groups; using a Z alpha in 1.65 and Z beta in 1.645, with a non-inferiority margin of 0.6; resulting in 98 subjects per group.

After obtaining the informed consent, patients will be randomized accordingly to their CD4+ T cell count (less or more than 50 cells/mm3 and assigned to each group:

* Group A or Conventional Steroids use (CoSt).patients will receive 21 days of steroid treatment.
* Group B or Shortened Steroids use (SSt). Subjects with moderate PCP will receive 8 days of steroids and subjects with severe PCP 14 days of steroids.

The equivalent prednisone doses of systemic steroids will be recorded, as well as the duration of their administration since it could be modified according to the criteria of the treating physicians; demographic data, the start date of ART (Antiretroviral Therapy), and the presence of other opportunistic, nosocomial and co-infections will also be recorded.

The laboratory data that will be recorded at the time of diagnostic suspicion of PCP will be: CD4+ T cell count, HIV viral load, lactate dehydrogenase (LDH), C-reactive protein (PCRe), pAO2, Da-aO2.

Once the patient has been discharged, the patient will be scheduled to continue ambulatory, conventional follow-up at 90, 180 and 360 days after starting the ART and to evaluate secondary outcomes.

Once 50% of the sample size has completed 30 days of follow-up, a preliminary analysis will be conducted to assess safety and efficacy; if differences in the mortality are observed, the study will be terminated.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* To have a gasometry at the admission that confirms moderate or severe PCP.
* Patients receiving trimethoprim / sulfamethoxazole in doses of 15 to 20 mg / kg per day from the first 24 hours after admission.
* Patients who have begun adjuvant treatment with steroids in the first 48 hours after admission.
* No history of chronic pulmonary disease.
* APACHE at hospitalization less than 20 points.

Exclusion Criteria:

* Allergic to TMP/SMX, who have not tolerated desensitization.
* History of inflammatory, infectious, autoimmune or neoplastic diseases except Kaposi's sarcoma, which merit the chronic use of steroids.
* Pleural or pericardial effusion and meningitis from any cause.
* Septic shock not related to PCP.
* Subjects who during the hospitalization have been diagnosed with any neoplasia (except Kaposi´s sarcoma)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of Mortality at 30 days | 30 days
  To compare 30-day cumulative incidence of mortality in subjects with moderate and severe PCP and HIV infection in patients receiving the shortened steroid scheme or the conventional 21-day schedule.

SECONDARY OUTCOMES:
Cumulative incidence of Mortality at 90 days | 90 days
  To compare cumulative incidence of mortality in patients receiving the shortened steroid scheme or the conventional 21-day schedule, at 90 days
Cumulative incidence of mortality at 360 days | 360 days
  To compare mortality in patients receiving the shortened steroid scheme or the conventional 21-day schedule
Cumulative incidence of mortality by CMV pneumonitis | 360 days
  To compare cumulative incidence of mortality stratified by the CMV pneumonitis (yes or not) in patients receiving the shortened steroid scheme or the conventional 21-day schedule, at 360 days
Cumulative incidence of mortality by CD4+T cell count | 360 days
  To compare cumulative incidence of mortality stratified by the CD4+ T cell count (less of or more than 50 cells per mm3), in patients receiving the shortened steroid scheme or the conventional 21-day schedule
Cumulative incidence of mortality by PCP severity | 360 days
  To compare cumulative incidence of mortality stratified by the PCP severity (moderate or severe), according with the gasometric parameters (AIDSinfo), in patients receiving the shortened steroid scheme or the conventional 21-day schedule
Time of intubation | 90 days
  To compare the time of intubation expressed in days of intubation,in subjects receiving the shortened steroid scheme or the conventional 21-day schedule
Time of intubation stratified by PCP severity | 90 days
  To compare the time of intubation expressed in days of intubation, in patients receiving the shortened and conventional steroid scheme, stratified by the PCP severity (moderate or severe), according with the gasometric parameters (AIDSinfo)
Number of participants with ventilatory requirements, stratified by the CD4+ T cell count | 90 days
  To compare the ventilatory requirements expressed by need for reintubation or intubation during hospitalization, in patients receiving the shortened and conventional steroid scheme, stratified by the CD4+ T cell count (less or more than 50 cells per mm3).
Number of participants with ventilatory requirements stratified by the CMV coinfection | 90 days
  To compare the ventilatory requirements, expressed by need for reintubation, in patients receiving the shortened and conventional steroid scheme, stratified by the CMV coinfection (yes or not)
Media of arterial oxygenation | 90 days
  To compare the arterial oxygenation thresholds using the media of arterial partial pressure of oxygen (PaO2) in arterial blood gasometry, obtained at admission, and 21 days in subjects receiving the shortened and conventional steroid scheme
Media of arterial oxygenation, stratified by PCP severity | 90 days
  To compare the arterial oxygenation thresholds using the media of arterial partial pressure of oxygen (PaO2) in arterial blood gasometry, obtained at admission, and 21 days in subjects receiving the shortened and conventional steroid scheme, stratified by the PCP severity (moderate or severe)
Media of arterial oxygenation, stratified by CD4+ T cell Count | 90 days
  To compare the arterial oxygenation thresholds using the media of arterial partial pressure of oxygen (PaO2) in arterial blood gasometry, obtained at admission, and 21 days in subjects receiving the shortened and conventional steroid scheme, stratified by the CD4+ T cell count (less or more than 50 cells per mm3)
Media of arterial oxygenation, stratified by the CMV pneumonitis | 90 days
  To compare the arterial oxygenation thresholds using the media of arterial partial pressure of oxygen (PaO2) in arterial blood gasometry, obtained at admission, and 21 days in subjects receiving the shortened and conventional steroid scheme, stratified by the presence or absence of CMV pneumonitis
Pulmonary function | 360 days
  To compare the pulmonary function, expressed by the spirometric pattern (normal, or obstructive, or restrictive), in pre and post-bronchodilator spirometry at 360 days in patients receiving the shortened and conventional steroid scheme.
Pulmonary function changes | 360 days
  To compare the changes in the spirometry pattern (normal, or obstructive, or restrictive), between baseline and 360 days in subjects receiving the shortened and conventional steroid scheme.
Pulmonary function by spirometry, stratified by CD4+ T cell count | 360 days
  To compare the pulmonary function, expressed by the spirometric pattern (normal, or obstructive, or restrictive), in pre and post-bronchodilator spirometry, in patients receiving the shortened and conventional steroid scheme, stratified by the CD4+ T cell count (less or more than 50 cells per mm3)
Pulmonary function by spirometry, stratified by PCP severity | 360 days
  To compare the pulmonary function, expressed by the spirometric pattern (normal, or obstructive, or restrictive), in pre and post-bronchodilator spirometry, in patients receiving the shortened and conventional steroid scheme, stratified by the PCP severity (moderate or severe)
Pulmonary function by spirometry, stratified by CMV pneumonitis | 360 days
  To compare the pulmonary function, expressed by the spirometric pattern (normal, or obstructive, or restrictive), in pre and post-bronchodilator spirometry, in patients receiving the shortened and conventional steroid scheme, stratified by the presence or absence of CMV pneumonitis
Changes in diffusing lung capacity of carbon monoxide | 360 days
  To compare the changes in the diffusing lung capacity of carbon monoxide (DLCO) in patients receiving the shortened and conventional steroid scheme
Changes in diffusing lung capacity of carbon monoxide by CMV coinfection | 360 days
  To compare the changes in the diffusing lung capacity of carbon monoxide (DLCO) in patients receiving the shortened and conventional steroid scheme, stratified by the CMV coinfection
Changes in diffusing lung capacity of carbon monoxide by the PCP severity | 360 days
  To compare the changes in the diffusing lung capacity of carbon monoxide (DLCO) in patients receiving the shortened and conventional steroid scheme, stratified by the PCP severity
Changes in diffusing lung capacity of carbon monoxide by CD4+ cell count | 360 days
  To compare the changes in the diffusing lung capacity of carbon monoxide (DLCO) in patients receiving the shortened and conventional steroid scheme, stratified by the CD4+ T cell count less or more than 50 cells per mm3
IRIS | 360 days
  Compare the cumulative incidence of IRIS associated with herpes virus infection 1, 2, 3, and 8, in patients receiving the shortened and conventional steroid scheme
Herpes virus dynamic | 90 days
  Measure the replication of herpes virus with the plasma viral load of Epstein-Barr Virus (EBV), Cytomegalovirus (CMV) and human herpes-virus 8 (HHV8) in blood

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Reyes-Teran, M.D., Principal Investigator — Instituto Nacional de Enfermedades Respiratorias
Locations (1):
- Centro de Investigacion en Enfermedades Infecciosas, México, Mexico

IPD SHARING:
Plan to Share IPD: No